CLINICAL TRIAL: NCT02449382
Title: To Effect and Safety of Continuous Venovenous Hemofiltration (CVVH) Versus Conventional Treatment for Acute Severe Hypernatremia in Critical Ill Patients: A Randomized Clinical Trial
Brief Title: Continuous Venovenous Hemofiltration Versus Conventional Treatment for Acute Severe Hypernatremia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, M.D., Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVVH-Na-002
Record Dates: First submitted 2015-05-11; First posted 2015-05-20 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Hypernatremia; Critically Ill
Keywords: continuous venovenous hemofiltration; conventional treatment; mortality; acute severe hypernatremia
MeSH Terms: conditions — Hypernatremia; Critical Illness | interventions — Continuous Renal Replacement Therapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous venovenous hemofiltration (Active Comparator): CVVH was mainly determined by the differences of sodium concentration between serum and replacement fluid. The rate of decline serum sodium could be real-time adjusted using different-sodium-concentration replacement fluid according to the updated serum sodium concentration.
  Interventions: Procedure: continuous venovenous hemofiltration
- Control group (Active Comparator): Treatment of hypernatremia is correction of water deficit.
  Interventions: Drug: Control group

INTERVENTIONS:
Procedure: continuous venovenous hemofiltration — If the serum sodium concentration >150mmol/L, When filter occurred clotting, replace the filter to CVVH treatment
  Other Names: continuous renal replacement therapy
  Arms: continuous venovenous hemofiltration
Drug: Control group — If the serum sodium concentration ≤150mmol/L, When filter occurred clotting, as the end of treatment.
  Other Names: standard treatments
  Arms: Control group

SUMMARY:
The patients with severe hypernatremia who received conventional treatment are often undertreated. Continuous venovenous hemofiltration (CVVH) can effectively remove solute or water from circulation system. Several case reports demonstrated that CVVH could effectively decrease serum sodium concentration of the patients with severe hypernatremia. The use of CVVH for acute severe hypernatremia in critically ill patients could improve patient survival by effectively decreasing the serum sodium concentration to a normal level.

DETAILED DESCRIPTION:
Date collection:

1. Demographic (gender, age, race, weight, history of drug allergy, complicating diseases, drug combination and combination therapy)
2. CVVH treatment (time, blood vessel, blood flow, replacement fluid flow, the type and dose of anticoagulant, limited to the test group)
3. Vital signs (blood pressure, heart rate, respiratory frequency, body temperature)
4. Severity of disease
5. General treatment (Vasoactive drugs, mechanical ventilation, diuretic, steroid hormones) 6.24 hours input 7.24 hour output

8.Daily sodium intake 9.Adverse events were confirmed 10.Laboratory date: Routine blood test Blood biochemical Blood gas analysis Blood electrolyte Plasma osmotic pressure Urine osmotic pressure Plasma osmotic pressure Urinary electrolyte excretion fraction

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Acute severe hypernatremia(increasing of serum sodium levels from normal levels to ≥160 mmol/L within 48 hours)
3. ICU patients

Exclusion Criteria:

1. Hypovolemic hypernatremia fractional excretion of sodium <0.5% and Urea/Creatinine >40 receiving diuretics: Urea/Creatinine >40, No edema.
2. Acute kidney injure network III
3. End-stage renal disease Hemodialysis or peritoneal dialysis
4. K+>6.5mmol/L The drug is difficult to treat hyperkalemia
5. Hydrogen ion concentration<7.2 The drug is difficult to treat metabolic acidosis
6. Acute pulmonary edema
7. Systolic blood pressure <90 mmHg vasoactive drugs in the treatment of systolic blood pressure less than 90 mmHg
8. The heparin or low molecular allergic patients
9. HIV positive patients
10. Pregnant women or lactational pregnancy women
11. Suspected tuberculosis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
7-day all cause mortality | 7days

SECONDARY OUTCOMES:
Glasgow Coma score changes | 3 days
  On the third day of the Glasgow Coma score minus baseline of the Glasgow Coma score
Sequential Organ Failure Assessment score changes | 3 days
  On the third day of the Sequential Organ Failure Assessment score minus baseline of the Sequential Organ Failure Assessment score
Acute Physiology and Chronic Health Evaluation II score changes | 3 days
  On the third day of the Acute Physiology and Chronic Health Evaluation II score minus baseline of the Acute Physiology and Chronic Health Evaluation II score
The average reduce rate of serum sodium | 3 days
  The average reduce rate of serum sodium was calculated as following: (serum sodium concentration before treatment (mmol/L) - serum sodium concentration after treatment (mmol/L)) / time after treatment (hours)
24-hour correction of hypernatremia | 24-hour
  Twenty-four-hour correction of hypernatremia was defined as the reduction of serum sodium concentration to ≤145 mmol/L within 24 hours after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shiren Sun, M.D., Principal Investigator — the First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- Xijing Hospital of Nephrology, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Huang C, Zhang P, Du R, Li Y, Yu Y, Zhou M, Jing R, Li L, Zheng Y, Wang H, Liu H, He L, Sun S. Treatment of acute hypernatremia in severely burned patients using continuous veno-venous hemofiltration with gradient sodium replacement fluid: a report of nine cases. Intensive Care Med. 2013 Aug;39(8):1495-6. doi: 10.1007/s00134-013-2933-9. Epub 2013 May 8. No abstract available. PMID 23653182